CLINICAL TRIAL: NCT03420703
Title: The Effect of Erector Spinae Plane Block on Postoperative Pain Following Laparoscopic Cholecystectomy: A Randomized Controlled Study
Brief Title: Erector Spinae Plane Block for Postoperative Analgesia for Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Can AKSU, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-349
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Pain
Keywords: erector spinae plane block; laparoscopic cholecystectomy; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block group (Active Comparator): Erector espine plane block will be administrated to this group. An intravenous patient controlled analgesia device will be given to the patients postoperatively
  Interventions: Other: erector spinae plane block; Device: Intravenous morphine patient controlled analgesia device
- control group (Sham Comparator): An intravenous patient controlled analgesia device will be given to the patients postoperatively
  Interventions: Device: Intravenous morphine patient controlled analgesia device

INTERVENTIONS:
Other: erector spinae plane block — ultrasound guided erector spinae plane block will be administered to this group.
  Arms: Block group
Device: Intravenous morphine patient controlled analgesia device — Intravenous morphine patient controlled analgesia device will be given to the patients postoperatively and 24 hour morphine consumption will be recorded

SUMMARY:
Erector Spinae Plane Block is a newly defined regional anesthesia technique. Its use for many indications has been identified by case reports in the literature. As the investigators have considered that erector spinae plane block could be efficacious for providing postoperative analgesia in laparoscopic cholecystectomy, the investigators have implemented application of this blockade into practice at the clinic. Main purpose of this study is to evaluate the analgesic effect of ultrasound guided erector spinae block in laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* 25 - 75 years of age
* ASA I - II
* Undergoing elective laparoscopic cholecystectomy

Exclusion Criteria:

* obesity
* ASA III - IV
* infection of the skin at the site of needle puncture area
* patients with known allergies to any of the study drugs
* coagulopathy
* recent use of analgesic drugs

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-02-24 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
24h morphine consumption | for postoperative 24 hour
  morphine consumptions for both group will be recorded

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | 24 hour
  PONV after surgery was questioned
Pain | 24h
  Numeric rating scales were recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Hospital, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided